CLINICAL TRIAL: NCT03239886
Title: Imatinib Discontinuation in Patients With Chronic Myeloid Leukemia Chronic Phase With Sustained MR4log
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15418
Record Dates: First submitted 2017-05-15; First posted 2017-08-04 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2017-05

CONDITIONS: Leukemia, Myeloid, Chronic-Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Intervention Model Description: single-arm study; all patients will discontinue imatinib (intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Discontinuation (Experimental): All subjects will discontinue imatinib
  Interventions: Other: imatinib discontinuation

INTERVENTIONS:
Other: imatinib discontinuation — imatinib discontinuation

SUMMARY:
This study will evaluate the proportion of subjects with chronic myeloid leukemia chronic phase that sustain major molecular response after imatinib discontinuation. To be eligible for this protocol, the subject must have received imatinib as first line regiment for at least 3 years with sustained molecular response of 4log (RM4log) or higher for one year.

DETAILED DESCRIPTION:
Patients will be followed for 2 years, with molecular monitoring, every month in the first year and then every 2 months. Imatinib will be restarted if the major molecular response (RM3log) is lost during the study or if the subject withdraw the informed consenting.

The primary objective is to measure the number of subject that sustain the major molecular response (RM3log or BCR-ABL level below 0.1%) after 2 years of follow-up.

BCR: breakpoint cluster region

ABL: abelson murine leukemia

RM3log: major molecular response, BCR-ABL level below 0.1% (IS)

ELIGIBILITY:
Inclusion Criteria:

* Chronic myeloid leukemia chronic-phase, defined by the World Health Organization criteria
* Treatment with imatinib for at least 36 months
* BCR-ABL levels below 0,01% (IS) or MR4log in the last 12 months

Exclusion Criteria:

* Previous allogeneic stem cell transplantation
* Previous treatment with dasatinib, nilotinib, bosutinib or ponatinib
* Imatinib dose escalation at any time, due to loss or inadequate response
* BCR-ABL mutation

IS: International Scale

MR4log: molecular response of 4log or <0,1% (IS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects that remain with RM3log after imatinib discontinuation | 24 months
  Number of subjects that sustain BCR-ABL level below 0,1% after 24 months of follow up.

SECONDARY OUTCOMES:
Number of subjects that recover MR3log after imatinib reintroduction | 6 months
  In the population that do not sustain BCR-ABL below 0,1% during the study, the time to recover the response after imatinib reintroduction will be measured
Analysis of immunological profile of all subjects | 24 months
  Study of lymphocytes population by flow cytometry, including NK and T population
Safety and tolerability of imatinib discontinuation | 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Pesquisa Clínica da Hematologia do HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seguro FS, Maciel FVR, Santos FM, Abdo ANR, Pereira TDM, Nardinelli L, Rocha V, Bendit I. MR 4log and low levels of NK cells are associated with higher molecular relapse after imatinib discontinuation: Results of a prospective trial. Leuk Res. 2021 Feb;101:106516. doi: 10.1016/j.leukres.2021.106516. Epub 2021 Jan 21. PMID 33517185